CLINICAL TRIAL: NCT02798471
Title: A Phase 3, Open-label, Randomized, Multi-center, Controlled Trial to Evaluate the Pharmacokinetics and Pharmacodynamics of Edoxaban and to Compare the Efficacy and Safety of Edoxaban With Standard of Care Anticoagulant Therapy in Pediatric Subjects From Birth to Less Than 18 Years of Age With Confirmed Venous Thromboembolism (VTE)
Brief Title: Hokusai Study in Pediatric Patients With Confirmed Venous Thromboembolism (VTE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DU176b-D-U312; 2016-000991-49 (EudraCT Number); CTRI/2018/01/011249 (Registry Identifier: Clinical Trials Registry - India (CTRI)); NCT02798471 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2016-05-11; First posted 2016-06-14 (Estimated); Results first posted 2023-03-06 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Venous Thromboembolism (VTE); Pulmonary Embolism; Deep Vein Thrombosis (DVT)
Keywords: Pediatric; Venous thrombolism; Pulmonary embolism
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism; Venous Thrombosis | interventions — edoxaban; Standard of Care; Warfarin; Heparin; Enoxaparin; Fondaparinux

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental): Edoxaban treatment will be dispensed to the participant on a monthly visit schedule.
  Edoxaban will be started orally at the age/weight/renal function appropriate dose, depending on the results of the ongoing U157 study (NCT02303431) for the Treatment Period.
  Interventions: Drug: Edoxaban
- Standard of Care (Experimental): Standard of Care (SOC) treatment will be dispensed to the participant on a monthly visit schedule.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Edoxaban — 15 or 30 mg tablets for participants 12 years of age to <18, and 60 mg edoxaban suspension for oral administration to participants under 12 years of age
  Arms: Edoxaban
Drug: Standard of Care — Standard of care could include low molecular weight heparin (LMWH), vitamin K antagonist (VKA), or synthetic pentasaccharide (SP) Xa inhibitors.
  Other Names: Warfarin/heparin; Enoxaparin; Fondaparinux
  Arms: Standard of Care

SUMMARY:
This is an event driven Phase 3, prospective, randomized, open-label, blinded endpoint evaluation (PROBE) parallel group study in subjects with confirmed VTE. This study is designed to evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of edoxaban and to compare the efficacy and safety of edoxaban against standard of care in pediatric subjects with confirmed VTE.

DETAILED DESCRIPTION:
The objective is to demonstrate the non-inferiority of edoxaban to standard of care (SOC; including low molecular weight heparin (LMWH), vitamin K antagonist (VKA), or synthetic pentasaccharide (SP) Xa inhibitors) in the treatment and secondary prevention of VTE in pediatric subjects with regard to the composite efficacy endpoint (ie, symptomatic recurrent VTE, death as result of VTE, and no change or extension of thrombotic burden) during the first 3-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female pediatric subjects between birth (defined as 38 weeks gestational age) and less than 18 years of age at the time of consent.
2. Pediatric subjects with the presence of documented VTE confirmed by appropriate diagnostic imaging and requiring anticoagulant therapy for at least 90 days.
3. Subjects must have received at least 5 days of heparin therapy prior to randomization to treat the newly identified index VTE. In addition, prior to being randomized to edoxaban or SOC, subjects initially treated with VKA are recommended to have an international normalized ratio (INR) < 2.0.
4. Subject and/or parent(s)/legal guardian(s) or legally acceptable representative is informed and provides signed consent for the child to participate in the study.
5. Female subjects who have menarche must test negative for pregnancy at Screening and must consent to avoid becoming pregnant by using an approved contraception method throughout the study.

Exclusion Criteria:

1. Subjects with active bleeding or high risk of bleeding contraindicating treatment with LMWH, SP Xa inhibitors, VKAs, or direct oral anticoagulants (DOACs; identified high risk of bleeding during prior experimental administration of DOACs).
2. Subjects who have been or are being treated with thrombolytic agents, thrombectomy or insertion of a caval filter for the newly identified index VTE.
3. Administration of antiplatelet therapy is contraindicated in both arms except for low dose aspirin defined as 1-5 mg/Kg/day with maximum of 100 mg/day.
4. Administration of rifampin is prohibited during the study and subjects on concomitant use of rifampin are excluded.
5. Subjects with hepatic disease associated with coagulopathy leading to a clinically relevant bleeding risk (aPTT > 50 seconds or international normalized ratio [INR] > 2.0 not related to anticoagulation therapy) or alanine aminotransferase (ALT) > 5 × the upper limit of normal (ULN) or total bilirubin > 2 × ULN with direct bilirubin > 20% of the total at Screening Visit.
6. Subjects with glomerular filtration rate (GFR) < 30% of normal for age and size as determined by the Schwartz formula.
7. Subjects with stage 2 hypertension defined as blood pressure (BP) systolic and/or diastolic confirmed > 99th percentile + 5 mmHg.
8. Subject with thrombocytopenia < 50 × 109/L at Screening Visit. Subjects with a history of heparin-induced thrombocytopenia may be enrolled in the study at the Investigator's discretion.
9. Life expectancy less than the expected study treatment duration (3 months).
10. Subjects who are known to be pregnant or breastfeeding.
11. Subjects with any condition that, as judged by the Investigator, would place the subject at increased risk of harm if he/she participated in the study, including contraindicated medications.
12. Subjects who participated in another clinical study or treated with an experimental therapy with less than a 30 day washout period prior to identifying the qualifying index VTE.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (140):
- United States (22):
  - Banner University Medical Center, Tucson, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Medical Center CAR, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Spectrum Health Helen DeVos Children's Hospital Grand Rapids, Grand Rapids, Michigan
  - Children's Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University North Carolina- Chapel Hill, Chapel Hill, North Carolina
  - Levine Children's Hospital Charlotte, Charlotte, North Carolina
  - The Presbyterian Hospital, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Le Bonheur Childrens Hospital, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital Italiano Regional del Sur, Buenos Aires
  - Sanatorio Allende, Córdoba
- Brazil (16):
  - Hospital Erasto Gaertner - Liga Paranaense de Combate ao Câncer, Curitiba, Paraná
  - IMIP - Instituto de Medicina Integral Professor Fernando Figueira, Pernambuco, Recife
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Instituto de Cardiologia do Rio Grande do Sul, Pôrto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos - Fundação Pio XII, Barretos, São Paulo
  - Centro de Hematologia e Hemoterapia - Hemocentro de Campinas - UNICAMP, Campinas, São Paulo
  - Centro Multidisciplinar de Estudos Clínicos - CEMEC, Santo André, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Hospital Samaritano, São Paulo
  - Hospital da Luz Amico Saude LTDA, São Paulo
  - Hospital Infantil Pequeno Príncipe, São Paulo
  - GRAACC - Grupo de Apoio ao Adolescente e à Criança com Câncer, São Paulo
  - UNIFESP - Universidade Federal de São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - HMCG - Hospital e Maternidade Dr. Christovão da Gama, São Paulo
- Bulgaria (4):
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MHAT - "National Heart Hospital" EAD, Sofia
  - MHAT 'Tokuda Hospital Sofia', EAD, Sofia
  - Medical Center for Specialized Ambulatory Medical Assistance for Children's Diseases, Sofia
- Canada (3):
  - Edmonton Clinic Health Academy, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - McMaster Children's Hospital, Hamilton, Ontario
- Chile (2):
  - Hospital El Carmen Dr. Luis Valentin Ferrada, Maipú
  - Clinica Las Condes, Santiago
- Croatia (4):
  - Clinical Hospital Centre Rijeka, Rijeka
  - General Hospital Zadar, Zadar
  - Children's Hospital Zagreb, Zagreb
  - University Hospital Centre Zagreb, University of Zagreb School of Medicine, Zagreb
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - CTC Hodonin s.r.o., Hodonín
  - Dětská klinika Fakultní nemocnice, Hradec Králové
  - University Hospital Pilsen, CZ, Pilsen
- Ålborg Universitetshospital, Aalborg, Denmark
- Hospital Nacional de Niños Benjamín Bloom, San Salvador, Salvador, El Salvador
- France (7):
  - Clinical Hospital Centre Cavale Blanche BREST, Brest, Finistere
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hôpital des enfants, CHU Toulouse, Toulouse, Haute Garonne
  - CHU Rennes - Hopital Sud, Rennes, Ille Et Vilaine
  - CHU Angers - Hôpital Hôtel Dieu, Angers
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - CHU Arnaud de Villeneuve, Montpellier
- Germany (2):
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Charite - Campus Virchow-Klinikum, Berlin
- Guatemala (2):
  - Unidad de Cirugía Cardiovascular de Guatemala (UNICAR), Guatemala City
  - Unidad Nacional de Oncología Pediátrica (UNOP), Guatemala City
- Hungary (4):
  - Semmelweis University 2nd Department of Pediatrics, Budapest
  - Central Hospital of Southern Pest - National Institute of Hematology and Infectious Diseases, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - University of Szeged, Department of Pediatrics, Szeged
- India (9):
  - Shree Krishna Hospital & Medical Research Centre, H M Patel Centre for Medical Care and Education, Karamsad, Gujarat
  - Nirmal Hospital, Surat, Gujarat
  - Jain Institute of Vascular Sciences, Bangalore, Karnataka
  - M. S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Government Medical College and Hospital, Nagpur, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Christian Medical College, Ludhiana, Punjab
  - Institute of Child Health, Kolkata, West Bengal
  - Indraprastha Apollo Hospitals, Delhi
- Israel (4):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah ein Kerem, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
- Strathmore University Medical Centre, Nairobi, Kenya
- Lebanon (3):
  - American University of Beirut Medical Center, Beirut
  - Saint George University Hospital Medical Center, Beirut
  - Hotel Dieu de France Hospital, Beirut
- Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan, Malaysia
- Erasmus MC Sophia, Rotterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- Panama (2):
  - INDICASAT AIP Site 7871, Panama City
  - INDICASAT AIP Site 7872, Panama City
- Portugal (4):
  - Hospital de Braga, Braga
  - Hospital da Senhora da Oliveira, Guimarães
  - Centro Hospitalar de Lisboa Central, E.P.E. - Hospital de Santa Marta, Lisbon
  - Centro Hospitalar de Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
- S.C Centrul Clinic Mediquest S.R.L, Sângeorgiu de Mureş, Romania
- Russia (2):
  - FSBI of Science "Kirov Scientific and Research Institute of Hematology and Blood Transfusion, FMBA", Kirov
  - Russian Scientific Center of Radiology and Nuclear Medicine of Ministry of Health of Russian Federation, Department of Pediatric Oncology, Moscow
- Serbia (2):
  - Mother and Child Health Care Institute of Serbia "Dr. Vukan Cupic", Belgrade
  - Clinical Center Kragujevac, Kragujevac
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's And Children's Hospital, Singapore
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Araba, Vitoria-Gasteiz, Álava
- Taiwan (5):
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital, Taipei
- Thailand (6):
  - Ramathibodi Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Chiang Mai University Hospital, Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (10):
  - Cukurova University Faculty of Medicine Balcali Hospital Pediatry Department, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Çocuk Sağlığı Ve Hastalıkları Hematoloji Onkoloji Eğitim Araştırma Hastanesi, Ankara
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Yeditepe University Oncology Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Izmir Tepecik Training and Research Hospital, Izmir
  - Izmir Dr. Behcet Uz Cocuk Hastaliklari ve Cerrahisi Egitim ve Arastirma Hastanesi, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Mersin University Health Research and Practice Hospital, Mersin
- Ukraine (3):
  - Regional Children's Clinical Hospital, Dnipro
  - CI of Healthcare Regional Children CH Gastroenterology Center Kharkiv NMU, Kharkiv
  - Children City Clinical Hospital, Poltava

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 290 participants who met all inclusion criteria and no exclusion criteria were randomized to receive either edoxaban or standard of care treatment; 286 patients received at least 1 dose of study drug (modified intent-to-treat population).
Groups:
- Edoxaban: Pediatric patients who were randomized to edoxaban treatment. Edoxaban was administered as 15 or 30 mg tablets for participants 12 years of age to <18, and 60 mg edoxaban suspension for oral administration to participants under 12 years of age.
- Standard of Care: Pediatric patients who were randomized to standard of care (SOC) treatment. Standard of care may have included low molecular weight heparin (LMWH), vitamin K antagonist (VKA), or synthetic pentasaccharide (SP) Xa inhibitors.
Period: Overall Study
Arm/Group | Edoxaban | Standard of Care
Started | 147 | 143
Modified Intent-to-Treat Population | 145 | 141
Completed | 128 (Due to data entry error, 1 additional patient included in this count was counted as both a study completer and as discontinued from the study; however, this patient was only included in the completer data.) | 119
Not Completed | 19 | 24
Not completed — Adverse Event | 7 | 2
Not completed — Physician Decision | 3 | 7
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 5 | 3
Not completed — Subject withdrew consent | 0 | 6
Not completed — Data entry error (reported as study completion and study discontinuation) | 2 | 0
Not completed — Randomized, but not treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics were reported in the Randomized Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Standard of Care | Total
Number analyzed (Participants) | 147 | 143 | 290
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 147 | 143 | 290
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (5.99) | 11.1 (6.03) | 11.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 70 | 140
  Male | 77 | 73 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 24 | 26 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 10 | 19
  White | 93 | 87 | 180
  More than one race | 15 | 8 | 23
  Unknown or Not Reported | 5 | 11 | 16
Region of Enrollment [Number; unit: participants]
  Singapore | 2 | 4 | 6
  United States | 24 | 17 | 41
  Czechia | 8 | 5 | 13
  Malaysia | 1 | 2 | 3
  Thailand | 7 | 8 | 15
  Portugal | 3 | 7 | 10
  Russia | 1 | 1 | 2
  Netherlands | 3 | 3 | 6
  South Korea | 6 | 3 | 9
  El Salvador | 5 | 0 | 5
  Panama | 1 | 0 | 1
  Brazil | 4 | 7 | 11
  Guatemala | 5 | 4 | 9
  Bulgaria | 3 | 1 | 4
  Chile | 1 | 1 | 2
  France | 1 | 4 | 5
  Croatia | 5 | 1 | 6
  Hungary | 12 | 11 | 23
  Ukraine | 4 | 0 | 4
  India | 3 | 5 | 8
  Spain | 4 | 6 | 10
  Lebanon | 4 | 5 | 9
  Canada | 4 | 9 | 13
  Turkey | 13 | 17 | 30
  Norway | 2 | 3 | 5
  Taiwan | 5 | 3 | 8
  Israel | 6 | 7 | 13
  Germany | 5 | 3 | 8
  Colombia | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Recurrent Venous Thromboembolism During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: Diagnosis of recurrent venous thromboembolism (VTE) requires the confirmation by diagnostic imaging and at least one of the symptoms of VTE from such areas as lower or upper extremity, catheter related thrombosis, pulmonary embolism, or sinovenous thrombosis.
Time Frame: Randomization to Month 3
Population: Symptomatic recurrent VTE was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 5 | 2
Statistical Analysis 1: Comparison: Edoxaban vs Standard of Care; Statistical analysis for the composite primary efficacy endpoint; Test type: Non-Inferiority — The edoxaban-to-comparator hazard ratio will be computed with 95% confidence interval (CI) (two-sided) based on this model. Edoxaban will be considered non-inferior to comparator if the upper limit of the 95% CI is ≤1.5; p = 0.9694, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.594 to 1.719]

2. Primary Outcome: Number of Participants Who Died as a Result of VTE During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: Death from venous thromboembolism (VTE) is based on objective diagnostic testing, autopsy or death which cannot be attributed to documented cause for which VTE cannot be ruled out.
Time Frame: Randomization to Month 3
Population: Death was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Pulmonary embolism (PE) with or without deep vein thrombosis (DVT) | 0 | 1
  Fatal PE | 0 | 0
  Non-fatal PE | 0 | 1
  Deep vein thrombosis (DVT) only | 5 | 1
  Fatal DVT | 0 | 0
  Non-fatal DVT | 4 | 0
  Unexplained death which VTE cannot be ruled out | 1 | 1

3. Primary Outcome: Number of Participants With No Change or Extension of Thrombotic Burden During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: No change or extension of thrombotic burden as assessed by quantitative diagnostic imaging of the index qualifying VTE thrombus at baseline and at Month 3. Imaging criteria for VTE included: - Abnormal compression ultrasonography where compression had been normal or, if non-compressible during screening, an increase in diameter of the thrombus during full compression; - An extension of the echogenic intra-luminal thrombus or absence of flow in the central venous system on Doppler ultrasonography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect, or an extension of non-visualization of veins in the presence of a sudden cut-off on venography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect on computed tomography angiogram (CTA).
Time Frame: Randomization to Month 3
Population: Change in thrombotic burden was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 21 | 29

4. Secondary Outcome: Number of Participants With Symptomatic Recurrent Venous Thromboembolism During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: as for outcome 1
Time Frame: From randomization up to Month 12
Population: Symptomatic VTE was assessed in the modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 7 | 2

5. Secondary Outcome: Number of Participants With Symptomatic Recurrent VTE During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Individual Component of Primary Efficacy Endpoint)
Description: as for outcome 1
Time Frame: Randomization to Month 3
Population: Symptomatic recurrent VTE was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Symptomatic VTE | 4 | 1
  Pulmonary embolism (PE) with or without deep vein thrombosis (DVT) | 0 | 1
  Deep vein thrombosis (DVT) only | 4 | 0

6. Secondary Outcome: Number of Participants Who Died as a Result of VTE During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: as for outcome 2
Time Frame: From randomization up to Month 12
Population: Death was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Pulmonary embolism (PE) with or without deep vein thrombosis (DVT) | 1 | 1
  Fatal PE | 0 | 0
  Non-fatal PE | 1 | 1
  Deep vein thrombosis (DVT) only | 6 | 1
  Fatal DVT | 0 | 0
  Non-fatal DVT | 5 | 0
  Unexplained death which VTE cannot be ruled out | 1 | 1

7. Secondary Outcome: Number of Participants Who Died as a Result of VTE During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Individual Component of Primary Efficacy Endpoint)
Description: as for outcome 2
Time Frame: Randomization to Month 3
Population: Death was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Death as a result of VTE | 1 | 1
  Unexplained death which VTE cannot be ruled out | 1 | 1

8. Secondary Outcome: Number of Participants With No Change or Extension of Thrombotic Burden During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: No change or extension of thrombotic burden as assessed by quantitative diagnostic imaging of the index qualifying VTE thrombus. Imaging criteria for VTE included: - Abnormal compression ultrasonography where compression had been normal or, if non-compressible during screening, an increase in diameter of the thrombus during full compression; - An extension of the echogenic intra-luminal thrombus or absence of flow in the central venous system on Doppler ultrasonography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect, or an extension of non-visualization of veins in the presence of a sudden cut-off on venography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect on computed tomography angiogram (CTA).
Time Frame: From randomization up to Month 12
Population: Change in thrombotic burden was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 35 | 47

9. Secondary Outcome: Number of Participants With Adjudicated Individual Component of Primary Efficacy Endpoints During the Main Treatment Period Following Edoxaban or Standard of Care Treatment
Description: Diagnosis of recurrent VTE requires the confirmation imaging and ≥1 symptom of VTE. Death from VTE is based on diagnostic testing, autopsy or death which cannot be attributed to documented cause for which VTE cannot be ruled out. No change or extension of thrombotic burden (quantitative diagnostic imaging) of the index qualifying VTE thrombus. Imaging criteria for VTE: - Abnormal compression ultrasonography where compression had been normal or, if non-compressible during screening, an increase in diameter of the thrombus during full compression; - An extension of the echogenic intra-luminal thrombus or absence of flow in the central venous system on Doppler ultrasonography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect, or an extension of non-visualization of veins in the presence of a sudden cut-off on venography. - An extension of an intraluminal filling defect, or a new intraluminal filling defect on computed tomography angiogram (CTA).
Time Frame: Randomization to Month 3
Population: Change in thrombotic burden was assessed in the modified intent-to-treat population (mITT).
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Symptomatic recurrent VTE | 4 | 1
  PE with or without DVT | 0 | 1
  DVT only | 4 | 0
  Death as a result of VTE | 1 | 1
  Unexplained death which VTE cannot be ruled out | 1 | 1
  No change or extension of thrombotic burden | 21 | 29

10. Secondary Outcome: Number of Participants Reporting Adjudicated All-Cause Mortality During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated)
Description: All-cause mortality is defined as death due to any cause. Adjudicated data are reported for overall all-cause mortality, all-cause mortality by the primary cause of death, and primary cause of death further described by additional specifications.
Time Frame: From randomization up to Month 12
Population: All-cause mortality was assessed in the modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Participants with adjudicated all-cause mortality during treatment period | 2 | 3
  Participants with adjudicated all-cause mortality occurring after treatment period | 1 | 0
  Venous thromboembolism (VTE)-related death | 1 | 1
  Venous thromboembolism (VTE)-related death: Unexplained death which VTE cannot be ruled out | 1 | 1
  Other known causes of death | 1 | 2
  Other known causes of death: Cancer | 0 | 1
  Other known causes of death: Infectious disease | 0 | 1
  Other known causes of death: Other | 1 | 0

11. Secondary Outcome: Number of Participants With Deep Vein Thrombosis, Catheter-related Thrombosis, Sino-venous Thrombosis, and Pulmonary Embolism During the Main, Extension, and Overall Treatment Periods Following Edoxaban or Standard of Care Treatment
Description: Deep vein thrombosis was assessed by ultrasonography or magnetic resonance venography (MRV), catheter-related thrombosis was assessed by ultrasonography or echocardiography, sino-venous thrombosis was assessed by brain MRI, and pulmonary embolism was assessed by nuclear ventilation/perfusion (V/Q) scanning.
Time Frame: From randomization up to Month 12
Population: Deep vein thrombosis, catheter-related thrombosis, sino-venous thrombosis, and pulmonary embolism were assessed in the modified intent-to-treat (mITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants
  Main Treatment: Participants with DVT only | 4 | 0
  Main Treatment: Participants with catheter-related thrombosis | 1 | 0
  Main Treatment: Participants with cerebral sino-venous DVT thrombosis | 0 | 0
  Main Treatment: Participants with PE with or without DVT | 0 | 1
  Extension Treatment: Participants with DVT | 1 | 0
  Extension Treatment: Participants with catheter-related thrombosis | 0 | 0
  Extension Treatment: Participants with sino-venous DVT thrombosis | 1 | 0
  Extension Treatment: Participants with PE | 1 | 0
  Overall Treatment: Participants with DVT | 5 | 0
  Overall Treatment: Participants with catheter-related thrombosis | 1 | 0
  Overall Treatment: Participants with sino-venous DVT thrombosis | 1 | 0
  Overall Treatment: Participants with PE | 1 | 1

12. Secondary Outcome: Number of Participants With Major and Clinically Relevant Non-Major Bleeding Events (On Treatment) During the Main Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: Any bleeding event defined as major and clinically relevant non-major bleeding (CRNM) events was reported. Major bleeding was defined as defined as a composite of any of the following: fatal bleeding; and/or symptomatic bleeding in critical area or organ such as intracranial, intra-spinal, intraocular, retroperitoneal, intra-articular, pulmonary, or pericardial, or intramuscular with compartment syndrome; and/or bleeding that causes a decrease in hemoglobin of at least 2 g/dL or more, or leading to transfusion of the equivalent of two or more units of whole blood or red blood cells. CRNM was defined as acute or sub-acute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of the following: a hospital admission for bleeding; a physician-guided medical or surgical treatment for bleeding or a change in antithrombotic therapy (including interruption or discontinuation of study drug).
Time Frame: Randomization to Month 3
Population: Major and clinically relevant non-major bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 3 | 5

13. Secondary Outcome: Number of Participants With All Bleeding Events (On Treatment) During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: All bleeding events included major bleeding defined as a composite of any of the following: fatal bleeding; and/or symptomatic bleeding in critical area or organ such as intracranial, intra-spinal, intraocular, retroperitoneal, intra-articular, pulmonary, or pericardial, or intramuscular with compartment syndrome; and/or bleeding that causes a decrease in hemoglobin of at least 2 g/dL or more, or leading to transfusion of the equivalent of two or more units of whole blood or red blood cells (RBCs), clinically relevant non-major bleeding defined as acute or sub-acute clinically overt bleed that does not meet the criteria for a major bleed but prompts a clinical response, in that it leads to at least one of the following: a hospital admission for bleeding; a physician-guided medical or surgical treatment for bleeding or a change in antithrombotic therapy (including interruption or discontinuation of study drug), nuisance bleeding, or a combination of bleeding events.
Time Frame: From randomization up to Month 12
Population: All bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 25 | 24

14. Secondary Outcome: Number of Participants With Major and Clinically Relevant Non-Major Bleeding Events (On Treatment) During the Overall Treatment Period Following Edoxaban or Standard of Care Treatment (Adjudicated Composite)
Description: as for outcome 12
Time Frame: From randomization up to Month 12
Population: Major and clinically relevant non-major bleeding events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban | Standard of Care
Number analyzed (Participants) | 145 | 141
Participants | 8 | 5

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the date the Informed Consent Form was signed up to Month 12.
Arm/Group | Edoxaban | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/145 | 3/141
Serious Adverse Events (participants affected / at risk) | 44/145 | 37/141
Other Adverse Events (participants affected / at risk) | 51/145 | 46/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=145) | Standard of Care (N=141)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Sickle cell anemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 6
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Chronic granulomatous disease (Congenital, familial and genetic disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Medical device site rash (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Rhinovirus infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 4 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Stoma complication (Injury, poisoning and procedural complications) | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Lipoedema (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Anaplastic astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Idiopathic intracranial hypertension (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Cerebral venous sinus thrombosis (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 1
Psychiatric decompensation (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 1
Superior vena cava occlusion (Vascular disorders) | 1 | 0
Venoocclusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban (N=145) | Standard of Care (N=141)
Vomiting (Gastrointestinal disorders) | 16 | 9
Pyrexia (General disorders) | 12 | 11
Nasopharyngitis (Infections and infestations) | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 8
Headache (Nervous system disorders) | 20 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT02798471/Prot_SAP_000.pdf